CLINICAL TRIAL: NCT03198234
Title: Use of T-allo10 Cell Infusions Combined With Mismatched Related or Mismatched Unrelated Hematopoietic Stem Cell Transplantation (HSCT) for Hematologic Malignancies
Brief Title: Use of T-allo10 in Hematopoietic Stem Cell Transplantation (HSCT) for Blood Disorders
Acronym: T-allo10
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Roncarolo, Maria Grazia, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rajni Agarwal, Associate Professor of Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-38734; PEDSBMT297 (Other: OnCore); 5P01CA049605-30 (NIH)
Record Dates: First submitted 2017-04-11; First posted 2017-06-26 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: AML - Acute Myeloid Leukemia; MDS (Myelodysplastic Syndrome); Mixed Phenotype Acute Leukemia; NHL - Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma; ALL
Keywords: Pediatric; GvHD; Hematopoietic Stem Cell Transplantation; Stem Cells; Transplant; BMT - bone marrow transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Leukemia, Biphenotypic, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants will receive 1 X 10^6/kg (± 10%) T-allo10 cells infused intravenously on Day -1 (day before transplant)
  Interventions: Biological: T-allo10
- Cohort 2 (Experimental): Participants will receive 3 X 10^6/kg (± 10%) T-allo10 cells infused intravenously on Day -1 (day before transplant)
  Interventions: Biological: T-allo10
- Cohort 3 (Experimental): Participants will receive 9 X 10^6/kg (± 10%) T-allo10 cells infused intravenously on Day -1 (day before transplant)
  Interventions: Biological: T-allo10

INTERVENTIONS:
Biological: T-allo10 — The T-allo10 drug product consists of donor derived, host (patient) alloantigen hyporesponsive (anergic) CD4+ (cluster of differentiation 4) cells containing Type 1 regulatory T (Tr1) cells induced in vitro in the presence of IL-10 (interleukin-10), which are also defined as IL-10 anergized T cells. T-allo10 cell infusion is being developed to prevent acute Graft-versus-Host Disease (GvHD) and induce graft tolerance in patients with hematologic malignancies receiving mismatched related and unrelated unmanipulated hematopoietic stem cell transplant (HSCT).

SUMMARY:
A significant number of patients with hematologic malignancies need a hematopoietic stem cell transplant (HSCT) to be cured. Only about 50% of these patients have a fully matched donor, the remaining patients will require an HSCT from a mismatched related or unrelated donor. Almost 60% of these mismatched donor HSCTs will result in graft-versus-host disease (GvHD), which can cause significant morbidity and increased non-relapse mortality. GvHD is caused by the donor effector T cells present in the HSC graft that recognize and react against the mismatched patient's tissues.

Researchers and physicians at Lucile Packard Children's Hospital, Stanford are working to prevent GvHD after HSCT with a new clinical trial. The objective of this clinical program is to develop a cell therapy to prevent GvHD and induce graft tolerance in patients receiving mismatched unmanipulated donor HSCT. The cell therapy consists of a cell preparation from the same donor of the HSCT (T-allo10) containing T regulatory type 1 (Tr1) cells able to suppress allogenic (host-specific) responses, thus decreasing the incidence of GvHD.

This is the first trial of its kind in pediatric patients and is only available at Lucile Packard Children's Hospital, Stanford.

The purpose of this phase 1 study is to determine the safety and tolerability of a cell therapy, T-allo10, to prevent GvHD in patients receiving mismatched related or mismatched unrelated unmanipulated donor HSCT for hematologic malignancies.

DETAILED DESCRIPTION:
Patients ages 3-30 years, with hematologic malignancies undergoing mismatched related or unrelated donor transplant will receive conditioning chemotherapy with Total body radiation and cyclophosphamide, according to the standard procedure.

The investigators plan to infuse the donor T-allo10 product one day before HSCT so that the Tr1 cells contained within the T-allo10 product will be able to prevent anti-host alloreactivity of the T cells present within the unmanipulated HSC graft. Indeed, Tr1 cells best exert their suppressive activity at the time of effector T cell activation, occurring when the T cells present in the HSC graft will be transferred to the patient ; therefore, the investigators expect that the early infusion of T-allo10 cells will optimally modulate anti-host alloreactivity of the donor T cells and prevent GvHD.

Immunosuppression will also be administered at the time of HSCT.

Up to 27 eligible patients will be given the T-allo10 product sequentially in 3 escalating dose cohorts to determine the maximum tolerated dose (or the highest dose tested if no maximum tolerated dose is reached). Each cohort will begin by evaluating 3 patients. The patients in each cohort will be staggered by 28 days and each succeeding patient will be enrolled no sooner than the 29 day after the preceding patient's infusion of T-allo10.

* If no patient in a cohort develops a dose limiting toxicity (DLT) following infusion of the investigational cellular product, the investigators will start enrolling patients at the next higher cell dose after completing the 28-day safety evaluation of the 3rd patient in the dose cohort.
* If one out of 3 patients in a cohort has a DLT, 3 additional patients will be evaluated at the same dose level.
* If one out of 6 patients experiences a DLT, dose escalation will occur.
* If 2 out of ≤ 6 patients experience a DLT, dose escalation will cease and that dose will be designated the maximally administered dose.
* Up to three (3) additional patients will be entered at the next lowest dose level if only 3 patients were treated previously at that dose

ELIGIBILITY:
Inclusion Criteria:

1. Eligible diseases include:

   A. Acute Lymphoblastic Leukemia (B- or T-ALL)
   1. Complete Response (CR)1-ultra high risk features

      * Unfavorable cytogenetics
      * Hypodiploidy
      * Induction failure
      * Minimal Residual Disease (MRD) positive after consolidation
   2. CR-2:

      * Any of the high risk features listed in CR1
      * B-ALL: any relapse considered eligible for transplant
      * T- ALL
   3. CR-3-any

   B. Acute Myeloid Leukemia
   1. MRD >5% at day 22 induction 1
   2. MRD >0.1% after induction 2
   3. FLT/ITD with allelic ratio > 0.4 and MRD >0.1% at day 22 or 29 induction 1
   4. Translocation (6:9), (8:6), (16:21), monosomy 7, monosomy 5, 5q
   5. M7 with KMT2A rearrangements, inv(16)(p13.3q24.3) [CBFA2T3-GLIS2] or t(11;12)(p15;p13) [NUP98-KDM5A]
   6. AML in 2nd or subsequent CR
   7. Therapy related or Secondary AML
   8. Refractory anemia with excess blasts (RAEB)2

   C. Myelodysplastic syndrome D. Mixed Phenotype Acute Leukemia MRD>1% after consolidation E. Non-Hodgkin's lymphoma (NHL) or Hodgkin's lymphoma (HL) beyond first remission
2. Age ≥3 to ≤45 years old. Subjects 1 and 2 (in Cohort 1) will be ≥ 12 years old
3. Available mismatched related donor (mMRD) or mismatched unrelated donor (mMUD), Human leukocyte antigen (HLA) matched 8/10 or 9/10
4. Lansky (age <16) or Karnofsky (age ≥16) performance status ≥80%
5. Able and willing to provide written, signed informed consent (assent as appropriate)
6. Have adequate organ function defined as the following:

   * Serum Creatinine <1.5 X upper limit of normal (ULN) or 24-hour creatinine clearance >50 ml/min
   * Serum bilirubin ≤ 2 x ULN
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)

     ≤10 x ULN
   * Diffusion Capacity of the Lungs (DLCO) >60% predicted (in children, O2 saturation >92% on room air)
   * Left ventricular ejection fraction >45% (in children, shortening fraction >26%)
7. Male and female subjects of child bearing potential must agree to use an effective method of birth control to avoid pregnancy throughout the transplant procedure, while on immunosuppression, and if the subject experiences any chronic GvHD.

Exclusion Criteria:

1. Prior bone marrow or peripheral blood HSCT within the last 6 (six) months
2. HLA-matched related or unrelated donor available
3. Any active, uncontrolled infection at the time of enrollment
4. Pregnant or lactating females
5. Any severe concurrent disease which, in the judgement of the investigator, would place the patient at increased risk during participation in the study
6. Any subject with a history of significant renal, hepatic, pulmonary, or cardiac dysfunction or on treatment to support cardiac dysfunction
7. HIV positive
8. Non-cooperative behavior or non-compliance of the patient and/or of his/her family
9. Received another investigational agent within 30 days of enrollment
10. Patients with Down's syndrome

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajni Agarwal, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Participants receive 1 X 10^6/kg (± 10%) T-allo10 cells infused intravenously on Day -1 (day before transplant)
- Cohort 2: Participants receive 3 X 10^6/kg (± 10%) T-allo10 cells infused intravenously on Day -1 (day before transplant)
- Cohort 3: Participants receive 9 X 10^6/kg (± 10%) T-allo10 cells infused intravenously on Day -1 (day before transplant)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 3 | 2 | 0
Completed | 3 | 1 | 0
Not Completed | 0 | 1 | 0
Not completed — Relapse of primary disease | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Cohort 1 was completed, and Cohort 2 enrolled two participants before closing due to feasibility.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5
Diagnosis [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia (AML) | 2 | 2 | 4
  Acute Lymphoid Leukemia (ALL) | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment Emergent Adverse Events (TEAE)
Description: Number of participants experiencing TEAEs. Assessments of TEAE will include laboratory abnormalities, changes in vital signs, and changes in physical examination related to the infusion of T-allo10 cells in order to assess the tolerability of T-allo10.
Time Frame: Time of T-allo10 cell infusion until 28 days following the infusion.
Population: One participant who had no post-transplant data is excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 1
Participants | 1 | 0

2. Primary Outcome: Severity of Treatment Emergent Adverse Events (TEAE)
Description: Number of participants experiencing TEAEs related to infusion, by severity graded according to the CTCAE grading system, from grade 1 (least severe) to grade 5 (death). Assessments of TEAE will include laboratory abnormalities, changes in vital signs, and changes in physical examination following infusion of T-allo10 cells in order to assess the safety of T-allo10.
Time Frame: Time of T-allo10 cell infusion until 28 days following the infusion.
Population: One participant who had no post-transplant data is excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 1
Participants
  Grade 1 | 1 | 0
  >=Grade 2 | 0 | 0

3. Primary Outcome: Number of Participants Who Achieved Stem Cell Engraftment After Hematopoietic Stem Cell Transplant (HSCT).
Description: Stem cell engraftment is evaluated by clinical laboratory studies including absolute neutrophil count above 500/mm3 for three consecutive days, hematopoiesis at bone marrow examination, with cellularity >5 % and donor chimerism >90% by short tandem repeat (STR) analysis for the presence of donor cells, and minimal residual disease (MRD) assay < 0.1%.
Time Frame: +42 days post HSCT
Population: One participant who had no post-transplant data is excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 1
Participants | 3 | 1

4. Primary Outcome: Number of Successful T-allo10 Products Manufactured for Patients Enrolled
Description: Feasibility defined by the rate of successful manufacture of the T-allo10 product to satisfy the targeted dose level and meet the required release specifications. Number of products meeting specifications out of total products manufactured is reported.
Time Frame: By Day -2
Measure: Count of Units; unit: Products
Units Other Than Participants: Products
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 2
Number analyzed (Products) | 3 | 2
Products | 3 | 0

5. Secondary Outcome: Number of Participants Who Experienced Grade III and/or IV Acute GvHD
Description: The number of patients who experienced grade III and IV acute GvHD at Day +100 following infusion of Tallo10 cells, assessed using the Modified Keystone scale administered by an independent evaluator on study visits through Day +100
Time Frame: Study visits through Day +100
Population: One participant who had no post-transplant data is excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 1
Participants | 2 | 0

6. Other Pre Specified Outcome: Number of Patients Who Developed Chronic GvHD
Description: The number of participants who experienced chronic GvHD and severity will be assessed by an independent evaluator. Outcome is reported as the highest level of chronic GVHD reported.
Time Frame: After Day +100 through Day +365
Population: One participant who had no post-transplant data is excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 1
Participants
  Mild | 2 | 0
  Moderate | 1 | 1
  Severe | 0 | 0
  Overall Incidence | 3 | 1

7. Other Pre Specified Outcome: Number of Days to Reach Immune Reconstitution
Description: Immune reconstitution will be evaluated by clinical laboratory studies of CD3+ T cells, assessed by the number of days to reach >200/microliter CD3+ T cells.
Time Frame: Up to Day 365
Population: One participant who had no post-transplant data is excluded from analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 1
Days | 22 [21 to 28] | 56 [56 to 56]

8. Other Pre Specified Outcome: Number of Participants Who Experienced Disease Free Survival
Description: Disease free survival is defined as the absence of minimal residual disease in the bone marrow.
  The investigators will use bone marrow aspirate examination, minimal residual disease (MRD) assay, and donor chimerism by STR analysis to evaluate disease free survival.
Time Frame: At Day +365
Population: One participant who had no post-transplant data is excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 1
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were recorded up to 1 year post-transplant.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=2)
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Duodenal hematoma (Vascular disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Fever (General disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Viremia: RSV (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=2)
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1
Alanine aminotransferase increased (ALT) (Investigations) | 3 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
AML relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Aspartate aminotransferase increased (AST) (Investigations) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood in stool (Gastrointestinal disorders) | 0 | 1
Body aches (General disorders) | 0 | 1
Breakthrough bleeding (Reproductive system and breast disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholesterol high (Investigations) | 2 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cramps in legs (with bowel movement) (Investigations) | 1 | 0
Creatinine increased (Investigations) | 1 | 1
Cushingoid appearance (Endocrine disorders) | 1 | 0
D-dimer increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0
Elevated procalcitonin (Investigations) | 1 | 0
Enterocolitis infectious (C.difficile) (Infections and infestations) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Erythema (hairline) (Skin and subcutaneous tissue disorders) | 1 | 1
Eye infection (Infections and infestations) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Eyelid swelling (Eye disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Fever (General disorders) | 2 | 0
Fibrinogen decreased (Investigations) | 0 | 1
Flattened affect (Psychiatric disorders) | 1 | 0
Flushed face (Vascular disorders) | 1 | 0
Folliculitis (Skin and subcutaneous tissue disorders) | 1 | 1
Gingival bleeding (Blood and lymphatic system disorders) | 0 | 1
Gum swelling (Gastrointestinal disorders) | 1 | 0
GVHD: Chronic eyes (Immune system disorders) | 0 | 1
GVHD: Chronic GI (Immune system disorders) | 1 | 0
GVHD: Chronic Liver (Immune system disorders) | 0 | 1
GVHD: Chronic skin (Immune system disorders) | 2 | 1
GVHD: Acute GI (Immune system disorders) | 1 | 0
GVHD: Acute skin (Immune system disorders) | 2 | 0
Haptoglobin decreased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Hematuria (Renal and urinary disorders) | 1 | 1
High Blood Urea Nitrogen (BUN) (Metabolism and nutrition disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperchloremia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2
Hypoproteinemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased GGT (Investigations) | 1 | 1
Increased LDH (Investigations) | 2 | 1
Infusion-related reaction (General disorders) | 1 | 0
International normalized ratio (INR) increased (Investigations) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Intracranial hypertension (Nervous system disorders) | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 0
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lightheadedness (Nervous system disorders) | 1 | 0
Lip lesion (Gastrointestinal disorders) | 1 | 0
Low bicarbonate (Metabolism and nutrition disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Mild sensitivity to spicy foods (Gastrointestinal disorders) | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Oral pain (Gastrointestinal disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain: generalized (General disorders) | 1 | 0
Pain: gingival (Gastrointestinal disorders) | 1 | 0
Pain: neuropathic (Nervous system disorders) | 1 | 0
Pain: pelvic (Reproductive system and breast disorders) | 1 | 0
Pain: perianal (Reproductive system and breast disorders) | 1 | 0
Papulopustular rash (face) (Skin and subcutaneous tissue disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 0
Platelet count decreased (Investigations) | 3 | 2
Positive occult blood (Gastrointestinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash: Acneform (body) (Skin and subcutaneous tissue disorders) | 0 | 1
Rash: Acneform (face) (Skin and subcutaneous tissue disorders) | 0 | 1
Rash: Erythematous, lacy (extremities) (Skin and subcutaneous tissue disorders) | 1 | 0
Rash: Erythematous, lacy (trunk) (Skin and subcutaneous tissue disorders) | 1 | 0
Rash: Impetigo (Skin and subcutaneous tissue disorders) | 0 | 1
Rash: Maculo-papular (body) (Skin and subcutaneous tissue disorders) | 0 | 1
Rash: Maculo-papular (face) (Skin and subcutaneous tissue disorders) | 1 | 1
Redman syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin infection (Staphylococcus aureus) (Infections and infestations) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin redness (Skin and subcutaneous tissue disorders) | 2 | 0
Striae on arms (Skin and subcutaneous tissue disorders) | 1 | 0
Striae on legs (Skin and subcutaneous tissue disorders) | 1 | 0
Striae on trunk (Skin and subcutaneous tissue disorders) | 1 | 0
Systolic murmur (Cardiac disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Total lung capacity decreased (Infections and infestations) | 0 | 1
Upper airway congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viremia: Adenovirus (Infections and infestations) | 2 | 0
Viremia: Adenovirus (stool) (Infections and infestations) | 1 | 0
Viremia: CMV (Infections and infestations) | 3 | 1
Viremia: CMV (bone marrow) (Infections and infestations) | 0 | 1
Viremia: CMV (intestine) (Infections and infestations) | 1 | 0
Viremia: COVID-19 (Infections and infestations) | 0 | 1
Viremia: EBV (Infections and infestations) | 2 | 0
Viremia: HHV6 (Infections and infestations) | 3 | 1
Viremia: Parvovirus (Infections and infestations) | 1 | 0
Vitamin D deficiency (Investigations) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Watering eyes (Eye disorders) | 0 | 1
Weight loss (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 2 | 1
Wound infection (MSSA) (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination led to a small number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT03198234/Prot_SAP_000.pdf